CLINICAL TRIAL: NCT05984732
Title: Intergenerational Connections: Reminiscence and Digital Storytelling to Improve Social and Emotional Well-being of Older Adults With ADRD
Brief Title: Intergenerational Reminiscence and Digital Storytelling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Collaborators: Retirement Research Foundation (Other)
Responsible Party: Principal Investigator, Ling Xu, Associate Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: #2021-0206
Record Dates: First submitted 2023-07-14; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Alzheimer Disease
Keywords: ADRD; DST; reminiscence; older adult; young adult volunteer; RCT
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reminiscence with digital storytelling (Experimental): Older adults in the intervention group will receive 10 sessions of life-review or reminiscence discussion with the trained young adult volunteers (1-1.5 hours each week for 10 weeks). At the end of the study, they create a digital storybook based on their previous discussion.
  Interventions: Behavioral: Reminiscence with digital storytelling
- Social wellness with scrapbook or journal (Sham Comparator): Older adults in the control group will have general social wellness discussion with the young adult volunteers. At the end of the study, they will create a journal/scrapbook.
  Interventions: Behavioral: Social wellness with scrapbook or journal

INTERVENTIONS:
Behavioral: Reminiscence with digital storytelling — The older and young adult participants will be randomly assigned into the intervention (reminiscence) or control (social wellness) groups and then be randomly matched as dyads within each group. Older adults in the intervention group will receive 10 sessions of life-review with the trained young adult volunteers (1-1.5 hours each week for 10 weeks). During weeks 1-6, a life history interview will be carried out with different themes in each week: major turning points in life (W1), family history (W2), life/career accomplishments (W3), history of loves and hates (W4), stress experiences (W5), and meaning and purpose of life (W6). During weeks 7-10, the dyads will develop the DST together using tablets already owned by the UTA School of Social Work. The contents of sessions 7-10 will be structured as: outline/script, plan and storyboard (W7), film and record (W8), evaluate, integrate and finalize (W9), and publish/share (W10).
  Arms: Reminiscence with digital storytelling
Behavioral: Social wellness with scrapbook or journal — Older adults in the control group will have general social wellness discussion with the young adult volunteers, instead of structured reminiscence guidelines. The topics are: diet and health (week 1); exercise/activity and health (week 2); emotions and health (week 3); religious/spiritual practices and health (week 4); family/friend relationships and health (week 5); and social activities/engagement and health (week 6). For weeks 7-10, instead of DST, the young adult volunteer will work with the older adult to create an unstructured, non-digital record of the social visit related to wellness in later life (e.g. wellness scrapbook/journal).
  Arms: Social wellness with scrapbook or journal

SUMMARY:
The goal of this clinical trial is to develop and test how reminiscence offered by trained young adult volunteers using a digital storytelling (DST) platform may help older persons with Alzheimer's disease and related dementias (ADRD) to improve their social and emotional well-being. The main questions it aims to answer are:

1. Whether is this reminiscence and DST based intervention effective in improving social and emotional well-being of older adults with ADRD?
2. Whether do young adult participants improve their social and emotional well-being as well as knowledge and attitudes towards aging after participating this study?

Older adult participants in the intervention group will receive 6 sessions of life-review with young adult volunteers and create a DST based on their life review discussion in the last 4 weeks. Older adult participants in the social wellness control group will receive 6 sessions of general talks with young adults and create a non-digital scrapbook or journal at week 7-10. Researchers will compare these two groups to see if participants in the intervention group benefit more on their well-being.

DETAILED DESCRIPTION:
Project Significance:

The number of persons aged 65 and older with Alzheimer's disease and related dementias (ADRD) is estimated to reach 7.1 million by 2025. Most older adults with ADRD live in the community and many of them live alone. There is growing concern about social isolation, loneliness, and diminished emotional well-being among persons with ADRD. Research suggests that reminiscence strategies combined with an intergenerational approach may yield significant social and mental health benefits for older adults. Recently, experts have recommended the production of a digital life story book as part of reminiscence. Reminiscence is typically implemented by trained professionals (e.g. social workers, nurses), however, there has been growing interest in using trained volunteers due to staffing shortages and the costs associated with reminiscence programs. The proposed study will develop and test how reminiscence offered by trained young adult volunteers using a digital storytelling (DST) platform may help older persons with ADRD to improve their social and emotional well-being. The proposed study is well-aligned with the RRF Foundation for Aging's mission to improve the quality of life for older people and also addresses a key research priority of RRF Foundation for Aging, social and intergenerational connectedness.

Project Goals and Objectives:

Goal 1: Quantitatively test the effectiveness of this intervention in improving social well-being of older adults with ADRD. The objectives are to: (1) provide a 10-session intervention with reminiscence and DST to older adults by trained young adult volunteers, and (2) test whether older adults report significant improvement in quality of life and/or a decline in loneliness after the intervention.

Goal 2: Quantitatively test the effectiveness of this intervention in improving emotional well-being of older adults with ADRD. The objectives are to: (1) provide a 10-session intervention with reminiscence and DST to older adults by trained young adult volunteers, and (2) test whether older adults report significant changes in affect and/or resilience after the intervention.

Goal 3: Quantitatively test attitudes towards aging of the young adult volunteers. The objectives are to: (1) offer opportunities for trained young adult volunteers to engage with older adults in the 10-session intervention, and (2) test changes of their attitudes towards aging after the intervention with surveys.

Goal 4: Quantitatively test knowledge and awareness of ADRD disease of the young adult volunteers. The objectives are to: (1) offer a three-hour training to the young adult volunteers before the intervention starts, which covers the biological aspects of ADRD and how to communicate and connect interpersonally to persons with ADRD, and (2) test changes in their reported knowledge and awareness of ADRD with surveys.

Goal 5: Qualitatively evaluate the usefulness of this intervention from perspectives of the dyads. The objectives are to: (1) explore and interpret the statistical results obtained in goals 1-2 through individual interviews with older adults who report the greatest and least changes in well-being and attitudes toward aging; and (3) examine dyads participants' perceptions of the intervention in terms of quality, benefits, and usefulness.

Methods:

Sampling and recruitment. Participants in this study will be older adults living in the community and youth participants who are currently enrolled as undergraduate or graduate students at one large university. Prior power analysis showed a total of 92 dyads are required to test the effectiveness of the proposed intervention. Older adults with ADRD will be recruited through a community partnership with Tarrant County Meals On Wheels. Recruitment of young adult volunteers will target student organizations that have established relationships with the faculty as well as through faculty teaching. All participant recruitment (i.e. older and younger adults) will occur through phone calls and/or Microsoft Teams.

Study design. The proposed project will conduct a randomized control trial to assess the effects of the intervention. The older and younger participants will be randomly matched as dyads. Subsequently, the matched dyads will be randomly assigned into the intervention or control groups. Data will be collected at baseline prior to the intervention, mid- intervention, at the end of the intervention, and 3 months after the intervention.

An explanatory sequential mixed methods design will be utilized involving first collecting and analyzing the quantitative survey data to identify subsamples of participants who report the greatest and least changes in outcome measures, and then conducting qualitative interview of these subsamples. Of the individuals with the highest 10% (n = 5) or lowest 10% (n = 5) of changes based on survey tests, we will conduct follow up qualitative interviews through phone calls/Microsoft Teams to capture the details of their perceptions of the intervention and present a more robust analysis, taking advantage of the strengths of both methods.

Intervention. Before the intervention starts, the young adult volunteers will be required to attend a group training. Subsequently, older adults in the intervention group will receive 10 sessions of life-review with young adult volunteers. During week 1-6, a life history interview will be carried out with different themes in each week: major turning points in life (W1), family history (W2), life/career accomplishments (W3), history of loves and hates (W4), experiences of suffering or stressful experiences (W5), and meaning and purpose of life (W6). Guidelines for conducting a life history interview will be prepared for the young adult volunteers based on the work of Watt and Cappeliez. After each session, the young adult participant will write a one-page summary and reflect on the interview to help prepare the subsequent DST. During weeks 7-10, the dyad participants will develop the DST together using a password protected, encrypted tablet provided by the university. The contents of sessions 7-10 will be structured as: outline/script, plan and storyboard (W7), film and record (W8), evaluate, integrate and finalize (W9), and publish/ share (W10). Telephone-based intervention will be conducted for this study.

Measurement and data analysis. The primary outcomes of the study will be social and emotional well-being of older adults, and the secondary outcomes are the benefits of young adult volunteers. For social well-being, quality of life is a relatively global and stable phenomenon that comprehensively measures people's psychosocial well-being, and will be measured by quality of life-Alzheimer's disease (QoL-AD). Loneliness represents the negative subjective experience of the inadequacy of social relationships and will be measured with the De Jong Gierveld Loneliness Scale. For emotional well-being, positive and negative affect have been used to describe affective, emotional components of subjective well-being. It will be measured by Positive and Negative Affect Schedule (PANAS). Resilience, as an important emotional well-being indicator, assesses one's ability to bounce back or adapt to stressful situations or crises and will be measured by the Brief Resilience Scale (BRS). For the young adult volunteers, attitude towards aging will be measured with the Fraboni Scale of Ageism (FSA). Knowledge and awareness of ADRD disease is measured by the Alzheimer's Disease Knowledge Scale (ADKS). For research goals 1 to 4, quantitative analysis of covariate-adjusted linear mixed models for repeated measures will be computed to compare the intervention and control groups over time on the major outcomes of older adults and youth volunteers. For research goal 5, conventional content analysis of qualitative interviews will be conducted.

Potential regional or national impact:

The study, if successful, will lead to a replicable intervention that will have the potential for broader implementation in additional regions through community partners such as Area Agencies on Aging and Meals On Wheels. The proposed evaluation activities will allow us to determine the applicability of intergenerational reminiscence with DST as an effective intervention for supporting the social and emotional needs of persons with ADRD. After further field testing, the intervention may be scaled up to be implemented as a tool of practice across universities and communities in the U.S. and with larger numbers of clients, thereby maximizing its impact as an intervention to strengthen the social and emotional well-being of older adults with ADRD.

ELIGIBILITY:
The inclusion criteria of the older adult participants are those who:

* are aged 65 years or older;
* have cognitive impairment measured by Ascertain Dementia 8 screening scale;
* have decisional capacity as measured by the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC) ;
* are not participating any other research protocol currently;
* can speak and understand English.

The exclusion criteria for older adults are:

* participating in another trial or intervention;
* have health issues that prevent them from participating in the study for 3 months;
* cannot commit to be available for the full 10 weeks of intervention.

The inclusion criteria for the young adult volunteers are:

* age 18-30 years old;
* currently enrolled as a student at UTA when the study is conducted;
* can commit to be available for the full 10 weeks of the intervention.

The exclusion criteria for the young adult volunteers are:

* not current UTA student in the time of the study;
* have health issues or limited availability that prevent them from participating for the entire 10 weeks of intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 206 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Quality of life of older adults | up to 6 months
  Older adults' quality of life will be measured using the Quality of Life-Alzheimer's Disease (QoL-AD). Thirteen items will be asked with each rated by a scale of 1-4 (poor, fair, good, or excellent). Sum scores will be calculated for final analysis with a potential range of 13-52. The higher the QoL-AD score, the better is the quality of life.
Affect of older adults | up to 6 months
  Positive affect (PA) and negative affect (NA) of older adults will be conducted with Positive and Negative Affect Schedule (PANAS). Ten positive and Ten negative emotions will be asked using a 5-point scale. Sum scores will be calculated with higher scores indicating more PA and NA respectively, with potential range of 10-50 for each sum score.
Resilience of older adults | up to 6 months
  Resilience of older adults will be measured using the Brief Resilience Scale (BRS). Six items will be asked and each item ranges from 1 (low resilience) to 5 (high resilience). Total scores will be calculated for final analysis with a potential range of 6-30. The higher the sum score, the more resilience of older adults.
Loneliness of older adults | up to 6 months
  Loneliness will be measured by the De Jong Gierveld Loneliness Scale. Six items will be asked, each is measured with a 5 Likert scale. High sum scores indicate great loneliness with a potential range of 6-30.

SECONDARY OUTCOMES:
Loneliness of young adult | up to 6 months
  Loneliness of young adult will be measured by De Jong Gierveld Loneliness Scale. Sum scores will be calculated with higher sum scores indicating more loneliness, with a potential range of 6-30.
Knowledge of ADRD | up to 6 months
  Young adults' knowledge of ADRD will be measured with the Alzheimer's Disease Knowledge Scale (ADKS). Thirty items will be asked as true or false. Total scores will be calculated for final analysis with a potential range of 0-30. Higher scores indicate more knowledge of ADRD.
Attitudes toward aging | up to 6 months
  Young adults;s attitudes toward aging will be measured with the Fraboni Scale of Ageism (FSA). Twenty nine statements will be raged based on a 4-point Likert scale. Higher sum scores indicate more ageism of young adults, with a potential range of 29-116.

OTHER OUTCOMES:
To qualitatively evaluate the usefulness of this intervention from the perspectives of the selected Dyads | interview will last for up to 60 minutes
  Follow-up qualitative interviews will be conducted to explore participants' overall experience with and perceptions about the intervention. On the basis of the results from the survey, the investigators will select participants who have the highest and lowest levels of changes in the loneliness outcomes for further qualitative interviews (10 dyads in total). Each generation's experiences, perspectives, challenges, and suggestions regarding this intervention will be asked during these in-depth interviews. Content analyses will be conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Arlington, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu L, Fields NL, Daniel KM, Cipher DJ, Troutman BA. Reminiscence and Digital Storytelling to Improve the Social and Emotional Well-Being of Older Adults With Alzheimer's Disease and Related Dementias: Protocol for a Mixed Methods Study Design and a Randomized Controlled Trial. JMIR Res Protoc. 2023 Sep 7;12:e49752. doi: 10.2196/49752. PMID 37676706